CLINICAL TRIAL: NCT03772093
Title: The Effectiveness of Short-term Massage Versus Trabert Current Therapy in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-I-002/418/2013
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Low Back Pain
Keywords: massage; low back pain; Trabert current; Ultra-Reiz current
MeSH Terms: conditions — Low Back Pain | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with manual massage therapy (Active Comparator): 30 patients were randomly assigned to massage therapy. The procedures were performed for ten days, with weekend break. Manual massage of lumbar area was performed by certified massage therapist with the typical course of the procedure. The technique was consisted of stroking, kneading, grinding, patting and shaking. The procedure lasted twenty minutes.
  Interventions: Other: Manual massage
- Patients with Trabert current therapy (Active Comparator): 30 patients were randomly assigned to Trabert current therapy. The Trabert current was administered by 143 frequency, time of 2 ms impulse, time of break 5 ms. The current was generated by Pulsotronic ST-6D device (ZAMED©). The electric pads were placed on the lumbar area, in the middle part of spine. The anode in the lower part, near to buttocks. The intensity of current was regulated between 15-25 mA. The time of procedure lasted fifteen minutes.
  Interventions: Device: Trabert current

INTERVENTIONS:
Device: Trabert current — Trabert current is an interrupted direct current of low frequency (143 Hz) applied via medium sized electrodes supported on a thick moist viscose sponge. These electrodes are placed near the spinal column along the thoracolumbar region. The electrodes are separated from each other by a distance of 3-4 cms.The current is passed through electrodes placed on the body. The intensity of the current is gradually increased short of pain. The feeling should be a pronounced but a comfortable 'tingling' sensation ('comfortably strong'). By doing this, the optimum current strength specific to the patient is found. The intensity of the current is slowly increased in the first few minutes as patients get used to the sensation. It is thought that this current provides pain relief, reduces muscle spasm and increases blood flow.
  Other Names: Ultra-Reiz current
  Arms: Patients with Trabert current therapy
Other: Manual massage — Therapeutic massage is the manipulation of the soft tissue of whole body areas to bring about generalised improvements in health.Massage is thought to work through a mechanical action and a reflex action. A mechanical action is created by moving the muscles and soft tissues of the body using pressure and stretching movement. This mechanical action is based on breaking up fibrous tissue and loosen stiff joints.It may help heal damaged muscle, stimulate circulation, clear waste products via the lymphatic system, boost the activity of the immune system, reduce pain and tension and induce a calming effect.
  Arms: Patients with manual massage therapy

SUMMARY:
Background: Low back pain (LBP) is still a frequent health problem. Recurrance of symptoms leads to high absence at work. It was proved in previous studies that low back manual massage has a significant impact on pain reduction. Trabert current (TC) is common physical modality used in rehabilitation of patients with LBP. The aim of study was to assess the effectiveness of manual massage in comparison to TC in patients with LBP.

Methods: Sixty patients with LBP were enrolled in to the study. In all patients discopathy and spondyloarthrosis were diagnosed. The subjects were randomly assigned to two groups: massage (I=30) and TC (II=30) therapy. The procedures were performed for ten days. Pain intensity was assessed by Numerical Rating Scale. Quality of life and the degree of disability were evaluated by Oswestry Disability Index and Roland-Morris Disability Questionnaire.

Results: In both groups pain reduction and functional improvement were observed after therapy. However, better results were noticed in group I.

ELIGIBILITY:
Inclusion Criteria:

* confirmed in X-ray spondyloarthrotic changes in lumbar area of spine
* pain of lumbar area lasting than 1 year

Exclusion Criteria:

* cardiac rythm disturbances
* cardiac pacemaker
* heart failure
* pulmonary embolism
* atherosclerosis
* neoplasmatic diseases
* skin lesions or purulent changes in the area of procedure
* pregnancy
* advanced osteoporosis
* spine fractures
* fever

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
pain intensity measured by NRS (numerical rating scale) | NRS was measured before and after 10 days massage and Trabert current therapy groups
  Numerical raitng scale (NRS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control. NRS is10-point scale, where 0=no pain and 10=worst possible pain.

SECONDARY OUTCOMES:
quality of life measured by Oswestry Disability Index (ODI) | ODI was measured before and after 10 days massage and Trabert current therapy groups
  is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

OTHER OUTCOMES:
quality of life measured by Roland-Morris Disability Questionnaire (RMDQ) | RMQ was measured before and after 10 days massage and Trabert current therapy groups
  RMDQ is designed to assess self-rated physical disability caused by low back pain.widely. The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore vary from 0 to 24. The questionnaire contains sentences that people have used to describe themselves when they suffer from back pain.

REFERENCES:
- [Background] Rahimi A, Vazini H, Alhani F, Anoosheh M. Relationship Between Low Back Pain With Quality of Life, Depression, Anxiety and Stress Among Emergency Medical Technicians. Trauma Mon. 2015 May;20(2):e18686. doi: 10.5812/traumamon.18686. Epub 2015 May 25. PMID 26290857
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Rajfur J, Pasternok M, Rajfur K, Walewicz K, Fras B, Bolach B, Dymarek R, Rosinczuk J, Halski T, Taradaj J. Efficacy of Selected Electrical Therapies on Chronic Low Back Pain: A Comparative Clinical Pilot Study. Med Sci Monit. 2017 Jan 7;23:85-100. doi: 10.12659/msm.899461. PMID 28062862
- [Background] Pop T, Austrup H, Preuss R, Niedzialek M, Zaniewska A, Sobolewski M, Dobrowolski T, Zwolinska J. Effect of TENS on pain relief in patients with degenerative disc disease in lumbosacral spine. Ortop Traumatol Rehabil. 2010 Jul-Aug;12(4):289-300. English, Polish. PMID 20876922
- [Background] Facci LM, Nowotny JP, Tormem F, Trevisani VF. Effects of transcutaneous electrical nerve stimulation (TENS) and interferential currents (IFC) in patients with nonspecific chronic low back pain: randomized clinical trial. Sao Paulo Med J. 2011;129(4):206-16. doi: 10.1590/s1516-31802011000400003. PMID 21971895
- [Background] Shipton EA. Physical Therapy Approaches in the Treatment of Low Back Pain. Pain Ther. 2018 Dec;7(2):127-137. doi: 10.1007/s40122-018-0105-x. Epub 2018 Sep 18. PMID 30229473
- [Background] Chou R, Deyo R, Friedly J, Skelly A, Hashimoto R, Weimer M, Fu R, Dana T, Kraegel P, Griffin J, Grusing S, Brodt ED. Nonpharmacologic Therapies for Low Back Pain: A Systematic Review for an American College of Physicians Clinical Practice Guideline. Ann Intern Med. 2017 Apr 4;166(7):493-505. doi: 10.7326/M16-2459. Epub 2017 Feb 14. PMID 28192793
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727
- [Background] Sayilir S, Yildizgoren MT. The medium-term effects of diadynamic currents in chronic low back pain; TENS versus diadynamic currents: A randomised, follow-up study. Complement Ther Clin Pract. 2017 Nov;29:16-19. doi: 10.1016/j.ctcp.2017.07.002. Epub 2017 Jul 29. PMID 29122255
- [Background] Bellido-Fernandez L, Jimenez-Rejano JJ, Chillon-Martinez R, Gomez-Benitez MA, De-La-Casa-Almeida M, Rebollo-Salas M. Corrigendum to "Effectiveness of Massage Therapy and Abdominal Hypopressive Gymnastics in Nonspecific Chronic Low Back Pain: A Randomized Controlled Pilot Study". Evid Based Complement Alternat Med. 2018 Sep 6;2018:3601984. doi: 10.1155/2018/3601984. eCollection 2018. PMID 30271453
- [Background] Furlan AD, Giraldo M, Baskwill A, Irvin E, Imamura M. Massage for low-back pain. Cochrane Database Syst Rev. 2015 Sep 1;2015(9):CD001929. doi: 10.1002/14651858.CD001929.pub3. PMID 26329399